CLINICAL TRIAL: NCT04061291
Title: A Cross-sectional Study to Explore the Relationship Between the Level of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2) as Measured Using a New Device (Inflammacheck™) Against Existing Measurements of Lung Disease and Inflammation in Patients With Asthma and COPD, and Healthy Volunteers.
Brief Title: Study to Explore the Relationship Between the Level of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2) as Measured Using a New Device Against Existing Measures of Lung Disease
Acronym: EXHALE 1A
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2017/120
Record Dates: First submitted 2019-05-03; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-05

CONDITIONS: Asthma; COPD Exacerbation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional, observational study of EBC H2O2 levels, as measured by a novel device, 'Inflammacheck™', and other markers of disease severity and symptom control in patients with Asthma and COPD and volunteers with no history of lung disease.

DETAILED DESCRIPTION:
Current tools for assessing airway inflammation and oxidative stress, such as fibre-optic bronchoscopy with bronchial wall biopsy and bronchial fluid lavage, are mostly invasive procedures that are not suitable for routine clinical practice or regular repeat sampling. Sample analysis requires a series of laboratory measurements and results can take over 24 hours to become available.

Induced sputum analysis is a semi-invasive means of assessing airway inflammation but is not always well tolerated by patients and again is not suitable for repeat sampling.

Non-invasive methods of measuring airway inflammation assess exhaled gases. Fractional exhaled Nitric Oxide (FeNO) measures eosinophilic airway inflammation. However, this test requires controlled exhalation for at least 6 seconds, making the test unsuitable for patients with impaired lung function, who are often not able to sustain this length of breath. Furthermore FeNO does not provide information about neutrophilic airway inflammation, a recognised component of steroid insensitive asthma and Chronic Obstructive Pulmonary Disease (COPD).

In contrast, measurement of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2) is performed during normal tidal breathing, and is well tolerated even in patients with severe airways obstruction and those unable to perform a consistent controlled exhalation. It is also not limited to inflammatory cell specific inflammation.

To date, the measurement of EBC H2O2 has been used as a research tool only, due to the complex multiple procedural steps required to deliver a result from the collected exhaled breath. Exhalation Technology Ltd. have now developed a novel, handheld device (Inflammacheck™) which can produce an immediate measurement of EBC H2O2 levels at the patients side. By detecting EBC H2O2 levels immediately, Inflammacheck™ could tell clinicians and patients the current level of global airway inflammation in a simple, effort independent manner. This could be used by clinicians to diagnose asthma and COPD, to determine a patient's phenotype and to guide correct and personalised treatment. It could also measure increased levels of airway inflammation that may indicate an exacerbation.

The 'Inflammacheck™' device now requires a study in a clinical setting to determine whether it can differentiate asthma and COPD from healthy, whether it can distinguish mild from severe disease and whether it can detect an acute exacerbation of these chronic respiratory conditions. The acceptability and ease of use of the device also needs to be assessed for both patients and clinicians.

ELIGIBILITY:
Inclusion Criteria:

* • Male or Female, aged ≥16 years.

  * A confirmed, clinician made diagnosis of asthma for ≥ 6months supported by evidence of any of the following;

    * Airflow variability, with a variability in FEV1 or Peak Expiratory Flow (PEF) of >20% across clinic visits within the preceding 5 years, with concomitant evidence of airflow obstruction (FEV1/FVC ratio <70% on spirometry);
    * Airway reversibility with an improvement in FEV1 by ≥12% or 200 ml after inhalation of 400 μg of salbutamol (or equivalent bronchodilator) via a metered dose inhaler and spacer within the preceding 5 years;
    * Airway hyper-responsiveness demonstrated by Methacholine challenge testing with a provocative concentration of Methacholine required to cause a 20% reduction in FEV1 (PC20) of ≤ 16mg/ml or equivalent test.
  * Mild Asthma defined as GINA steps 1 to 3
  * Severe asthma defined as GINA steps 4 or 5
  * OR a confirmed, clinician made diagnosis of COPD for ≥ 6months supported by spirometric evidence of fixed airflow limitation (post-bronchodilator ratio of FEV1/FVC <0.7).
  * OR no known history of lung disease (defined as no current clinical diagnosis of, or be receiving treatment for, a lung disease).
  * Willing and able to give informed consent for participation in the study.

Healthcare Professionals Inclusion Criteria:

* Assisted a minimum of 5 patients in performing the collection of EBC H2O2 levels using the 'Inflammacheck™' device during the study.
* Willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:

  * Existing co-morbidities that may prevent them from performing spirometry, FeNO or other study measurements (at the discretion of the clinical investigator).
  * Known lung, chest wall, neuromuscular, or cardiac disease or abnormality that would confound symptom scores and spirometry.
  * In the opinion of the clinical investigator, participant would not be able to perform any of the study procedures.
  * Unable to comprehend the study and provide informed consent, e.g. insufficient command of English in the absence of someone to adequately interpret.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three populations of adult patients (all aged ≥18yrs) will be invited to participate:
  1. Asthma patients (n=50, 25 mild, 25 severe)
  2. COPD patients (n=50, 25 mild - moderate, 25 severe - very severe)
  3. Comparator group (n=50) - Volunteers with no previous history of lung disease (our 'healthy' volunteers). These healthy volunteers will be recruited from the hospital staff. This will be facilitated by the hospital and research communications teams. Healthcare Professionals, who have assisted patients performing 'Inflammacheck™', alongside the standard respiratory tests of spirometry and FeNO, will be invited to participate in an experience outcome questionnaire at the end of the study.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2018-02-03 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
Level of exhaled breath condensate hydrogen peroxide (EBC H2O2), | 1 day study visit
  EBC H202 as measured by the by Inflammacheck™ sensor

SECONDARY OUTCOMES:
Quality of life (asthma specific) | 1 day study visit
  measured by asthma quality of life questionnaire
  * Disease severity ( measured by GINA Stage for asthma, GOLD Stage for COPD)
  * Disease control (ACQ (asthma))
Quality of life (COPD specific) | 1 day study visit
  COPD assessment test
  * Rating of whether test is acceptable to participant
  * Participant's perception of device using the self perception questionnaire
Safety outcome | 1 day study visit
  incidence of adverse events reported during the study procedures
Disease Severity Asthma | 1 day study visit
  measured by Global Initiative for Asthma
Disease Severity COPD | 1 day study visit
  measured by Global Initiative for Chronic Obstructive Lung Disease

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No